CLINICAL TRIAL: NCT03599648
Title: Testing the Efficacy of Mindfulness-Based Stress Reduction Combined With Behavioral Parent Training in Families With Preschoolers With Developmental Delay
Brief Title: The Pro-Parenting Study: Helping Parents Reduce Behavior Problems in Preschool Children With Developmental Delay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: Loma Linda University (Other)
Responsible Party: Principal Investigator, Laura Lee McIntyre, Professor & Dean, College of Education, University of Oregon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HD093667-01A1 (NIH)
Record Dates: First submitted 2018-07-11; First posted 2018-07-26 (Actual); Results first posted 2025-03-03 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Development Delay; Behavior Problem
Keywords: intervention; behavioral parent training; mindfulness-based stress reduction
MeSH Terms: conditions — Learning Disabilities; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BPT-E (Experimental): Behavioral parent training (BPT) plus a psychoeducation program.
  Includes a 10-week standard BPT, plus a 6-week psychoeducation program delivered prior to the standard BPT.
  Interventions: Behavioral: BPT-E
- BPT-M (Experimental): Behavioral parent training (BPT) plus mindfulness-based stress reduction (MBSR).
  Includes a 10-week standard BPT, plus a 6-week MBSR delivered prior to the standard BPT.
  Interventions: Behavioral: BPT-M
- Teachers (No Intervention): At each wave of data collection, caregivers in both conditions were asked to identify a teacher who could provide an evaluation of their child's behavior outside the home. Participating teachers completed a brief 2-page questionnaire about the child.

INTERVENTIONS:
Behavioral: BPT-M — Participants randomized to the BPT-M condition receive the Mindfulness-Based Stress Reduction (MBSR) intervention, followed by Behavioral Parent Training (BPT). The MBSR module includes six weekly 2.5 hour group sessions, 30-45 minutes of daily home practice guided by audio CDs, and an MBSR parent workbook. In the sessions, participants practice formal mindfulness exercises, and are provided instruction on stress physiology and using mindfulness for coping with stress in everyday life.
  The BPT component of the intervention includes 10 weekly sessions lasting 2.5 hours. Each session is structured around videotape vignettes and uses discussion, role-playing, modeling, and feedback to foster mastery of the material. Parents are given weekly homework assignments and practice their skills.
  Arms: BPT-M
Behavioral: BPT-E — Participants randomized to the BPT-E condition will received 6 weeks of a psychoeducation program followed by 10 weeks of the Behavioral Parent Training (BPT) used in both conditions. The psychoeducation module consists of 6 weekly 2.5-hour sessions, daily homework that includes monitoring progress on goals identified at the end of each session, and a workbook for parents of children with special needs that provides parents with information regarding their child's development, disability, and associated considerations. Each of the 6 weekly sessions includes a general topic for discussion. These include preparing for IEP meetings, navigating the regional center and developmental service agencies, communicating with teachers, advocacy, sibling issues, and community resources.
  Arms: BPT-E

SUMMARY:
The Pro-Parenting Study seeks to determine the added benefit of targeting both parenting stress and parent management strategies to more effectively reduce behavior problems among children with developmental delay (DD). Findings from this study will improve the scientific understanding of evidence-based interventions for behavior problems among children with DD and the mechanisms underlying therapeutic change.

DETAILED DESCRIPTION:
Behavior problems are a common and concerning challenge among children with developmental delay (DD). Approximately 50% of children with DD have a comorbid mental disorder or serious behavior problems- a prevalence three times as high as that found in typically developing youths. Behavioral parent training (BPT) is the gold-standard intervention for treating child behavior problems in typically developing children and in children with DD. However, high levels of parental stress are associated with reduced or no response to BPT for children with DD. Consequently, parental stress may attenuate the efficacy of the gold-standard, empirically supported treatment for behavior problems among children with DD. As such, parental stress is a critical point of intervention for improving both parent and child outcomes in families of children with DD. The purpose of this study is to quantify the therapeutic benefit of adding a parent stress-reduction intervention prior to delivering BPT in order to more effectively reduce child behavior problems, and to investigate the mechanisms through which intervention outcomes occur.

ELIGIBILITY:
Inclusion Criteria:

* Parent has a child ages 3 to 5 years with an agency-identified DD in one or more functional areas who is receiving early intervention or early childhood/ preschool special education through an individualized family service plan (IFSP) or individualized education plan (IEP);
* Parent reports elevated child behavior problems, as indicated by a T-score of 60 or above on the Total Problems scale of the Child Behavior Checklist;
* Parent reports elevated parenting stress, as indexed by a total score above the recommended cutoff at the 85th percentile on the Parenting Stress Index-4.

Exclusion Criteria:

* Parent screens positive for active psychosis, substance abuse, or suicidality;
* Parent is currently receiving any form of psychological or behavioral treatment at the time of referral; or
* The child has sensory impairments or nonambulatory conditions that would necessitate the need for significant modifications to the lab and home visit protocols.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 959 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura L McIntyre, PhD, Principal Investigator — University of Oregon
Locations (2):
- United States (2):
  - Loma Linda University, Loma Linda, California
  - University of Oregon, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1041 families were assessed for eligibility, and 779 were excluded (591 did not meet inclusion criteria, 43 refused to participate, and 145 were excluded for other reasons such as not completing screening, geographic reasons, or scheduling challenges). In the end, 262 families (i.e., caregiver + child) were randomized and assigned to an arm. Children's current teachers were also invited to participate at each wave. A total of 660 teachers were invited; 438 completed a survey.
Groups:
- BPT-E: Behavioral parent training (BPT) plus a psychoeducation program.
  Includes a 10-week standard BPT, plus a 6-week psychoeducation program delivered prior to the standard BPT.
  BPT-E: Participants randomized to the BPT-E condition will received 6 weeks of a psychoeducation program followed by 10 weeks of the Behavioral Parent Training (BPT) used in both conditions. The psychoeducation module consists of 6 weekly 2.5-hour sessions, daily homework that includes monitoring progress on goals identified at the end of each session, and a workbook for parents of children with special needs that provides parents with information regarding their child's development, disability, and associated considerations. Each of the 6 weekly sessions includes a general topic for discussion. These include preparing for IEP meetings, navigating the regional center and developmental service agencies, communicating with teachers, advocacy, sibling issues, and community resources.
- BPT-M: Behavioral parent training (BPT) plus mindfulness-based stress reduction (MBSR).
  Includes a 10-week standard BPT, plus a 6-week MBSR delivered prior to the standard BPT.
  BPT-M: Participants randomized to the BPT-M condition receive the Mindfulness-Based Stress Reduction (MBSR) intervention, followed by Behavioral Parent Training (BPT). The MBSR module includes six weekly 2.5 hour group sessions, 30-45 minutes of daily home practice guided by audio CDs, and an MBSR parent workbook. In the sessions, participants practice formal mindfulness exercises, and are provided instruction on stress physiology and using mindfulness for coping with stress in everyday life.
  The BPT component of the intervention includes 10 weekly sessions lasting 2.5 hours. Each session is structured around videotape vignettes and uses discussion, role-playing, modeling, and feedback to foster mastery of the material. Parents are given weekly homework assignments and practice their skills.
- Teachers: Caregivers in both conditions were asked to identify a teacher at each wave of data collection who could provide an evaluation of the child's behavior outside the home. Teacher participation was not longitudinal, meaning that different teachers provided evaluations at each wave of data collection.
Period: Overall Study
Arm/Group | BPT-E | BPT-M | Teachers
Started (131 caregivers provided baseline data about themselves and their child. 128 children participated in play tasks at baseline, and two additional children participated for the first time at follow-up but are included here as having "started" the study. 80 teachers completed surveys about children at baseline.) | 261 | 260 (131 caregivers provided baseline data about themselves and their child. 128 children participated in play tasks, and one additional child participated for the first time at follow-up but is included here as having "started" the study. 90 teachers completed surveys about children at baseline.) | 438 (Teacher participation in the study was not longitudinal. This number represents the total number of teachers who participated at any wave of data collection. 170 teachers completed a survey at baseline, 107 at the time of immediate follow-up, 72 at the time of 6-month follow-up, and 89 at the time of 12-month follow-up.)
Received Intervention as Assigned (107 caregivers) | 107 | 114 (114 caregivers) | 0
Completed Follow-up Immediately After Intervention (At the time of immediate follow-up, 98 caregivers provided data about themselves and their child. 88 children participated in play tasks. 50 teachers completed surveys about children.) | 186 | 192 (At the time of immediate follow-up, 100 caregivers provided data about themselves and their child. 92 children participated in play tasks, including one who did not participate at baseline. 57 teachers completed surveys about children.) | 0
Completed 6-month Follow-up (At the time of 6-month follow-up, 97 caregivers provided data about themselves and their child. 86 children participated in play tasks, including two who did not previously participate at baseline or immediate follow-up. 32 teachers completed surveys about children.) | 183 | 187 (At the time of 6-month follow-up, 96 caregivers provided data about themselves and their child. 91 children participated in play tasks. 40 teachers completed surveys about children.) | 0
Completed 12-month Follow-up (At the time of 12-month follow-up, 104 caregivers provided data about themselves and their child. 90 children participated in play tasks. 40 teachers completed surveys about children.) | 194 | 201 (105 caregivers, 96 children, 49 teachers At the time of 12-month follow-up, 105 caregivers provided data about themselves and their child. 96 children participated in play tasks. 49 teachers completed surveys about children.) | 0
Completed (This number represents 109 caregivers and 106 children who completed at least one wave of data collection after the intervention was over.) | 215 | 219 (This number represents 111 caregivers and 108 children who completed at least one wave of data collection after the intervention was over.) | 438
Not Completed | 46 | 41 | 0

BASELINE CHARACTERISTICS:
Population: At baseline,131 caregivers in each condition provided data for themselves and their children, and 128 children in each condition participated in observation/ play tasks. Three additional children engaged in play tasks at later waves and are included here as having "started" the study. The current teacher of each child was recruited at each wave, resulting in a total of 438 teachers providing data about students at some point during the study. 170 teachers completed surveys at baseline.
Groups:
- Teachers: Regardless of treatment condition to which parents were assigned, children's current teachers were invited to participate at each wave of data collection. Participating teachers completed a 2-page questionnaire about their participating student. Because children moved to different classrooms with different teachers throughout the study, different teachers reported on a given child at each wave.
- Total: Total of all reporting groups
Arm/Group | BPT-E | BPT-M | Teachers | Total
Number analyzed (Participants) | 261 | 260 | 438 | 959
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One caregiver in the BPT-M condition did not answer question.
  Child age was measured in years in the first cohort but months in later cohorts. Given that age was measured differently for the first cohort, their data are not included here to simplify reporting.
  Teacher age was measured with ranges rather than exact years. These data are included in a separate table.
  years
    Caregivers: number analyzed (Participants) | 131 | 130 | 0 | 261
    Caregivers | 37.31 (7.65) | 37.32 (7.64) |  | 37.31 (7.63)
    Children: number analyzed (Participants) | 105 | 104 | 0 | 209
    Children | 4.28 (0.85) | 4.32 (.88) |  | 4.30 (.86)
    Teachers: number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Customized [Count of Participants; unit: Participants] — Population: Parent, child, and teacher age were all measured slightly differently, and thus appear in different tables. Teacher age was measured with ranges rather than exact years and those data are reported here. Age and demographic data were only collected from 274 teachers.
  Participants
    18-25 years: number analyzed (Participants) | 0 | 0 | 274 | 274
    18-25 years |  |  | 29 | 29
    26-35 years: number analyzed (Participants) | 0 | 0 | 274 | 274
    26-35 years |  |  | 89 | 89
    36-45 years: number analyzed (Participants) | 0 | 0 | 274 | 274
    36-45 years |  |  | 65 | 65
    46-55 years: number analyzed (Participants) | 0 | 0 | 274 | 274
    46-55 years |  |  | 58 | 58
    56-65 years: number analyzed (Participants) | 0 | 0 | 274 | 274
    56-65 years |  |  | 29 | 29
    66 years and older: number analyzed (Participants) | 0 | 0 | 274 | 274
    66 years and older |  |  | 2 | 2
    prefer not to answer: number analyzed (Participants) | 0 | 0 | 274 | 274
    prefer not to answer |  |  | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Demographic data were only collected from 274 teachers.
  Participants
    Caregivers: number analyzed (Participants) | 131 | 131 | 0 | 262
    Caregivers: Female | 128 | 124 |  | 252
    Caregivers: Male | 3 | 7 |  | 10
    Children: number analyzed (Participants) | 130 | 129 | 0 | 259
    Children: Female | 51 | 40 |  | 91
    Children: Male | 79 | 89 |  | 168
    Teachers: number analyzed (Participants) | 0 | 0 | 274 | 274
    Teachers: Female |  |  | 258 | 258
    Teachers: Male |  |  | 16 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographic data were only collected from 274 teachers.
  Participants
    Caregivers: number analyzed (Participants) | 131 | 131 | 0 | 262
    Caregivers: Hispanic or Latino | 80 | 72 |  | 152
    Caregivers: Not Hispanic or Latino | 45 | 57 |  | 102
    Caregivers: Unknown or Not Reported | 6 | 2 |  | 8
    Children: number analyzed (Participants) | 130 | 129 | 0 | 259
    Children: Hispanic or Latino | 87 | 83 |  | 170
    Children: Not Hispanic or Latino | 38 | 44 |  | 82
    Children: Unknown or Not Reported | 5 | 2 |  | 7
    Teachers: number analyzed (Participants) | 0 | 0 | 274 | 274
    Teachers: Hispanic or Latino |  |  | 96 | 96
    Teachers: Not Hispanic or Latino |  |  | 178 | 178
    Teachers: Unknown or Not Reported |  |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Demographic data were only collected from 274 teachers.
  Participants
    Caregivers: number analyzed (Participants) | 131 | 131 | 0 | 262
    Caregivers: American Indian or Alaska Native | 0 | 0 |  | 0
    Caregivers: Asian | 5 | 2 |  | 7
    Caregivers: Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
    Caregivers: Black or African American | 8 | 9 |  | 17
    Caregivers: White | 25 | 34 |  | 59
    Caregivers: More than one race | 7 | 12 |  | 19
    Caregivers: Unknown or Not Reported | 86 | 74 |  | 160
    Children: number analyzed (Participants) | 130 | 129 | 0 | 259
    Children: American Indian or Alaska Native | 1 | 1 |  | 2
    Children: Asian | 3 | 2 |  | 5
    Children: Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
    Children: Black or African American | 7 | 12 |  | 19
    Children: White | 32 | 41 |  | 73
    Children: More than one race | 10 | 4 |  | 14
    Children: Unknown or Not Reported | 77 | 69 |  | 146
    Teachers: number analyzed (Participants) | 0 | 0 | 274 | 274
    Teachers: American Indian or Alaska Native | 0 | 0 | 2 | 2
    Teachers: Asian | 0 | 0 | 24 | 24
    Teachers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Teachers: Black or African American | 0 | 0 | 16 | 16
    Teachers: White | 0 | 0 | 122 | 122
    Teachers: More than one race | 0 | 0 | 15 | 15
    Teachers: Unknown or Not Reported | 0 | 0 | 95 | 95
Region of Enrollment [Number; unit: participants] — Population: At baseline, 131 caregivers in the BPT-E and 131 caregivers in the BPT-M conditions provided baseline data about themselves and their child. However, only 128 children in each condition participated in play/ observation tasks at baseline (i.e., N=259 in each condition). At later waves, 3 children (2 in BPT-E and 1 in BPT-M) who did not participate in play tasks at baseline chose to do so, resulting in N=261 in BPT-E (131 parents + 130 children) and N=260 in BPT-M (131 parents + 129 children).
  participants
    United States | 261 | 260 | 438 | 959

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Child Behavior Problems (Parent Report)
Description: Parents report on child behavior using the Child Behavior Checklist-Ages 1.5-5 years (Achenbach, 2000), a 99-item questionnaire that assesses behavioral problems in young children. Parents were asked to rate how accurately each item described their child's behavior over the past 2 months using a 3-pt scale (0=not true/ 1= somewhat or sometimes true/ 2= very true or often true). A Total Behavior Problems score was derived by taking the sum of all 99 items, with a possible range of 0-198. A high score indicates greater problem behavior.
Time Frame: baseline, immediately after 16-week intervention, 6 months, 12 months
Population: Number of participants differs between baseline and follow-up waves due to attrition (e.g., participants not returning follow up surveys).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BPT-E | BPT-M
Number analyzed (Participants) | 121 | 122
score on a scale
  Baseline | 73.60 (27.77) | 77.95 (26.99)
  Immediately after 16-week intervention: number analyzed (Participants) | 84 | 89
  Immediately after 16-week intervention | 71.49 (29.51) | 71.69 (30.40)
  6-month follow-up: number analyzed (Participants) | 82 | 84
  6-month follow-up | 67.85 (29.51) | 70.67 (33.17)
  12-month follow-up: number analyzed (Participants) | 92 | 96
  12-month follow-up | 66.48 (29.43) | 68.25 (31.39)
Statistical Analysis 1: Comparison: BPT-E; Test type: Superiority; p = .361, t-test, 2 sided — baseline versus immediately after 16-week BPT-E intervention
Statistical Analysis 2: Comparison: BPT-E; Test type: Superiority; p = .126, t-test, 2 sided — baseline versus 6 months after BPT-E intervention
Statistical Analysis 3: Comparison: BPT-E; Test type: Superiority; p = .000, t-test, 2 sided — baseline versus 12 months after BPT-E intervention
Statistical Analysis 4: Comparison: BPT-M; Test type: Superiority; p = .000, t-test, 2 sided — baseline versus immediately after 16 week BPT-M intervention
Statistical Analysis 5: Comparison: BPT-M; Test type: Superiority; p = .000, t-test, 2 sided — baseline versus 6 months after BPT-M intervention
Statistical Analysis 6: Comparison: BPT-M; Test type: Superiority; p = .000, t-test, 2 sided — baseline versus 12 months after BPT-M intervention

2. Secondary Outcome: Change From Baseline in Parenting Behavior (Parent Report)
Description: Parents report on their parenting behavior using the Parenting Practices Interview (The Incredible Years, 2015), a 73-item questionnaire with 7 summary scales. Parents were asked how often they engaged in various parenting practices when their child misbehaved, or their likelihood of responding with a certain parenting behavior in provided scenarios of negative child behavior. The Appropriate Discipline summary scale (12 items) was used in the present study. Scores ranged from 1 to 7. Higher scores indicate greater use of appropriate disciplinary practices.
Time Frame: baseline, immediately after 16-week intervention, 6 months, 12 months
Population: Number of participants differs between baseline and follow-up waves due to attrition (e.g., participants not returning follow-up surveys).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BPT-E | BPT-M
Number analyzed (Participants) | 122 | 118
score on a scale
  Baseline | 3.85 (1.21) | 3.90 (1.03)
  Immediately after 16-week intervention: number analyzed (Participants) | 86 | 91
  Immediately after 16-week intervention | 4.02 (0.92) | 4.12 (1.02)
  6-month follow-up: number analyzed (Participants) | 82 | 84
  6-month follow-up | 4.10 (1.04) | 4.13 (1.06)
  12-month follow-up: number analyzed (Participants) | 89 | 93
  12-month follow-up | 4.15 (0.94) | 4.10 (0.99)
Statistical Analysis 1: Comparison: BPT-E; Test type: Superiority; p = .035, t-test, 2 sided — Baseline versus immediately following 16-week BPT-E intervention
Statistical Analysis 2: Comparison: BPT-E; Test type: Superiority; p = .001, t-test, 2 sided — Baseline versus 6-months after BPT-E intervention
Statistical Analysis 3: Comparison: BPT-E; Test type: Superiority; p = .000, t-test, 2 sided — Baseline versus 12 months after BPT-E intervention
Statistical Analysis 4: Comparison: BPT-M; Test type: Superiority; p = .000, t-test, 2 sided — Baseline versus immediately after 16-week BPT-M intervention
Statistical Analysis 5: Comparison: BPT-M; Test type: Superiority; p = .000, t-test, 2 sided — Baseline versus 6 months after BPT-M intervention
Statistical Analysis 6: Comparison: BPT-M; Test type: Superiority; p = .000, t-test, 2 sided — Baseline versus 12 months after BPT-M intervention

3. Secondary Outcome: Change From Baseline in Parenting Stress (Parent Self-Report)
Description: Parents report on their parenting stress using the Parenting Stress Index-Fourth Edition, Short Form (PSI4-SF; Abidin, 1995). Parents were asked to indicate their agreement with 36 statements about their feelings on a 5 pt scale (strongly agree, agree, not sure, disagree, strongly disagree). A Total Stress Score was derived from responses to these items, and scores could range from 36-180. High scores indicate greater parenting stress.
Time Frame: baseline, immediately after 16-week intervention, 6 months, 12 months
Population: Number of participants differs between baseline and follow-up due to attrition (e.g., participants not returning follow-up surveys).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BPT-E | BPT-M
Number analyzed (Participants) | 128 | 129
score on a scale
  Baseline | 113.70 (20.01) | 115.28 (20.86)
  Immediately After 16-week Intervention: number analyzed (Participants) | 83 | 89
  Immediately After 16-week Intervention | 101.23 (21.73) | 100.10 (20.80)
  6-month Follow-up: number analyzed (Participants) | 83 | 85
  6-month Follow-up | 97.72 (25.08) | 96.89 (22.33)
  12-month Follow-up: number analyzed (Participants) | 91 | 97
  12-month Follow-up | 96.21 (20.73) | 94.93 (26.40)
Statistical Analysis 1: Comparison: BPT-E; Test type: Superiority; p = .000, t-test, 2 sided — Baseline versus immediately after 16-week BPT-E intervention
Statistical Analysis 2: Comparison: BPT-E; Test type: Superiority; p = .000, t-test, 2 sided — Baseline versus 6 months after BPT-E intervention
Statistical Analysis 3: Comparison: BPT-E; Test type: Superiority; p = .000, t-test, 2 sided — Baseline versus 12 months after BPT-E intervention
Statistical Analysis 4: Comparison: BPT-M; Test type: Superiority; p = .000, t-test, 2 sided — Baseline versus immediately after 16-week BPT-M intervention
Statistical Analysis 5: Comparison: BPT-M; Test type: Superiority; p = .000, t-test, 2 sided — Baseline versus 6 months after BPT-M intervention
Statistical Analysis 6: Comparison: BPT-M; Test type: Superiority; p = .000, t-test, 2 sided — baseline versus 12 months after BPT-M intervention

ADVERSE EVENTS:
Time Frame: Caregivers and children were monitored for adverse events over the study period (e.g., up to 24 months from baseline).
Description: Adverse event data were not collected from teachers.
Groups:
- Teachers: Caregivers in both conditions were asked to identify a teacher at each wave of data collection who could provide an evaluation of the child's behavior at school. Teacher participation was not longitudinal, meaning that different teachers provided evaluations at each wave of data collection.
  Adverse events data were not collected from teachers.
Arm/Group | BPT-E | BPT-M | Teachers
All-Cause Mortality (participants affected / at risk) | 0/261 | 0/260 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/261 | 0/260 | 0/0
Other Adverse Events (participants affected / at risk) | 0/261 | 0/260 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT03599648/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/48/NCT03599648/ICF_001.pdf